CLINICAL TRIAL: NCT05174988
Title: Reducing Postoperative Bleeding After Hysterectomy Via Independent Closure of Vaginal Cuff Angles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Steven Radtke, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E22006
Record Dates: First submitted 2021-11-05; First posted 2022-01-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Bleeding; Patient Satisfaction; Complications; Operative Time
Keywords: bleeding; hysterectomy; cuff; closure
MeSH Terms: conditions — Postoperative Hemorrhage; Patient Satisfaction; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angle stitch (Experimental): If the allocation corresponds to "Angle stitch", surgeon will use 0 polyglactin 910 suture on a tapered needle to place figure of 8 sutures on both (left and right) apexes. Knot tying technique (intra-corporeal vs extracorporeal) will be up to surgeon preference. After this is completed, barbed suture will be used to re-approximate the remainder of the vaginal cuff from right to left, backtracking once at the end for reinforcement.
  Interventions: Procedure: Angle stitch
- control (No Intervention): If the subject's group corresponds to "Control group", the surgeon will re-approximate the cuff in a standard fashion, using a running-barbed suture (2-0 V-LOC 90 with tapered needle), starting at the right apex, moving towards the left, and then back-tracking once to further reinforce the closure.

INTERVENTIONS:
Procedure: Angle stitch — Surgeon will use 0 polyglactin 910 suture on a tapered needle to place figure of 8 sutures on both (left and right) vaginal cuff apexes.
  Arms: Angle stitch

SUMMARY:
The investigators propose prospectively evaluating if adding separate sutures to the angles of the vaginal cuff before running barbed suture reduces the incidence of patient's perception of bleeding after surgery.

DETAILED DESCRIPTION:
Hysterectomy is the most common surgical procedure in the United States, with over 600,000 performed annually.1 There has been a dramatic improvement in expected postoperative course secondary to the advancement of minimally invasive gynecologic surgery.2 With the advent of laparoscopy and robotic surgery, even the most complex cases can be successfully performed via a minimally invasive approach. What used to be a major surgery that required a prolonged inpatient stay has become an outpatient procedure where patients are discharged home a few hours after the operation.3 Although the recovery period is shorter than in the past, there are still some postoperative complaints that are relatively common, and can impair quality of life. One of them is postoperative vaginal bleeding. Although this can be a sign of a more serious problem such as vaginal cuff dehiscence, the grand majority of times it is related to granulation tissue in the vaginal cuff that although may be self-limiting, can be bothersome and concerning to patients. Not only does this bleeding impair quality of life, but it's one of the most common reasons for emergency room visits after surgery. Multiple studies have shown that postoperative vaginal bleeding and return to the hospital significantly affect patient satisfaction. 4,5 Anecdotally, bleeding originates from granulation tissue at the angles of the closure, although there hasn't been any studies specifically investigating this. A common approach to laparoscopic cuff closure involves a running barbed suture, with or without separate closure of the lateral angles.6,7 Recently, laparoscopic closure of the vaginal cuff was found to be superior when compared to vaginal closure in terms of vaginal cuff dehiscence8. This RCT also evaluated vaginal cuff bleeding as a secondary outcome, but this was recorded as he presence of bleeding at 3 months after surgery. The closure technique in this study was a running non-barbed suture, without independent suturing of the angles. Although a running suture placed laparoscopically may provide adequate tensile strength throughout the cuff to promote healing, the tension at the corners may be less than at the center when using barbed suture, hence potentially increasing the risk of bleeding. Furthermore, the second angle may be more difficult to access when the remainder of the cuff is re-approximated.

The investigators propose prospectively evaluating if adding separate sutures to the angles of the vaginal cuff before running barbed suture reduces the incidence of patient's perception of bleeding after surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Pre-menopausal patients scheduled to undergo hysterectomy via laparoscopic/robotic approach for benign indications (Ages 18-60, who have had at least one menstrual cycle in the last year).

Exclusion Criteria:

* Patient's that incur in an intraoperative bowel or urologic injury during the hysterectomy that requires repair. If injury occurs after randomization (during vaginal cuff closure), this will be recorded and reviewed by the study's safety officer

  * Patients scheduled to undergo a concomitant vaginal procedure (Mid-urethral sling, anterior/posterior repair)
  * Patients scheduled to undergo pelvic floor repair (utero-sacral ligament suspension)
  * Patients with known preoperative malignancy
  * Patients in which a total hysterectomy is not completed

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only patients undergoing a hysterectomy are eligible
Enrollment: 117 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
pain quantification on 0-10 scale | 10-20 days post intervention
  Pelvic pain scale from 0-10 assessed at postoperative visit, with 10 representing worse pain imaginable, and 0 representing no pain
postoperative bleeding frequency | 10-20 days post intervention
  Survey regarding postoperative vaginal bleeding- only if they are experiencing bleeding (categorical including Daily | Most days | Infrequent
prolonged bleeding | 90-110 days after intervention
  yes or no if any vaginal bleeding in the last 2 weeks
postoperative bleeding volume | 10-20 days post intervention
  Survey regarding postoperative vaginal bleeding- only if they are experiencing bleeding (categorical including Only when using restroom| Spotting throughout day | More than spotting

SECONDARY OUTCOMES:
Pain with sex on a 0-10 scale | 90-110 days after intervention
  Subjective scoring per patient of pain during intercourse on a scale of 0-10, where 10 is worst pain imaginable and 0 is no pain.
ER visits | 90-110 days
  emergency department visits related to surgery (yes or no)
Physical functioningSF36 | 90-110 days
  Calculated score Result from SF-36 (Short form-36 health survey) Range 0-100, with 100 representing the maximum of each particular outcome)
PainSF36 | 90-110 days
  Calculated score Result from SF-36 (Short form-36 health survey) Range 0-100, with 100 representing the maximum of each particular outcome)
General healthSF36 | 90-110 days
  Calculated score Result from SF-36 (Short form-36 health survey) Range 0-100, with 100 representing the maximum of each particular outcome)
Role limitations due to physical healthSF36 | 90-110 days
  Calculated score Result from SF-36 (Short form-36 health survey) Range 0-100, with 100 representing the maximum of each particular outcome)
Operative time | During the surgery. Start time begins when first suture and sewing instruments are in abdomen with the intention of closing vaginal cuff. Stop time is when last suture pertaining to vaginal cuff closure/apex stitches is cut.
  Vaginal cuff closure time in minutes recorded during the surgery. Start time begins when first suture and sewing instruments are in abdomen with the intention of closing vaginal cuff. Stop time is when last suture pertaining to vaginal cuff closure/apex stitches is cut.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Radtke, MD, Principal Investigator — Texas Tech University Health and Sciences Center
Locations (1):
- Texas Tech University Health Scince Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT05174988/Prot_000.pdf